CLINICAL TRIAL: NCT04598113
Title: The Immediate Effect of Cervical Traction on Balance in Cervical Radiculopathy Patients: A Randomized Cross-over Trial)
Brief Title: Effect of Cervical Traction on Balance in Cervical Radiculopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Anis Jellad, Professor, University of Monastir
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CTB
Record Dates: First submitted 2020-09-30; First posted 2020-10-22 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Cervical Radiculopathy; Vertigo
Keywords: Cervical Radiculopathy; Vertigo; Traction; Balance Postural
MeSH Terms: conditions — Radiculopathy; Vertigo

STUDY DESIGN:
Intervention Model Description: Two interventions: Effective Traction (ET) and Sham Traction (ST) Two arms: Arm 1: Effective Traction/Sham Traction (ET than ST) and Arm 2: Sham Traction/Effective Traction (ST than ET) Wash out period = 1 week
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant is treated with the same traction devise in the two interventions with just a traction intensity difference.
  The care provider who manipulate the traction device can't be blinded to allocation The investigator (performing balance tests) is blinded to the intervention type The outcome assessor is blinded to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effective Traction/Sham Traction (Active Comparator): Group of patients treated firstly with Effective Traction then with Sham Traction
  Interventions: Device: Cervical Traction Device
- Sham Traction/Effective Traction (Sham Comparator): Group of patients treated firstly with Sham Traction then with Effective Traction
  Interventions: Device: Cervical Traction Device

INTERVENTIONS:
Device: Cervical Traction Device — While The patient is lie on the back his or her head is housed within the specific head portion of the device. The investigator inflate progressively the device using a valve and ensuring the patient's relaxation. The process of inflation is continued until the level of 12 Kg of pressure is reached. This maximum level of traction is maintained for 10 minutes then the process of deflation is started until the pressure decreased to 0 Kg. This maneuver is reproduced once again after 5 minutes of rest.
  The balance assessment using the force plate-from is done just before the intervention and 5 minutes after its end.

SUMMARY:
A cross-over randomized trial aiming to assess the immediate effect of cervical traction on balance disorders among patients with common cervical neuropathy. Authors hypothesized that as cervical traction alleviate radicular pain it may also improve patient balance disorders. Effective traction is compared to sham traction.

Main outcome measures are balance parameters (force platform).

DETAILED DESCRIPTION:
A cross-over randomized trial was designed to assess the immediate effect of cervical intermittent traction on balance disorders among patients diagnosed with common cervical neuropathy. The diagnosis is confirmed or made by a physical medicine and rehabilitation physician with 15 Y of experience treating musculoskeletal disorders especially cervical neuropathy. Enrolled patients are randomly assigned to one of two arms (1 or 2). Patients in arm 1 (Effective Traction/Sham Traction) are treated firstly with effective traction than one week later with sham traction. Patients in arm 2 (Sham Traction/Effective Traction) are treated firstly with sham traction than one week later with effective traction. At baseline the epidemiological parameters, the pain intensity (VAS), the grip strength, the functional status (NDI), the psychological distress (HAD), the Brief Best Test and the balance parameters (force platform) are assessed. The pain intensity, the grip strength and the balance parameters are assessed before and immediately after cervical traction for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cervical radiculopathy of greater than three months

Exclusion Criteria:

* History of surgery or bone-ligament damage to the cervical spine
* Neurological and/or rheumatic diseases involving the cervical spine or which may result in impaired balance
* Inner ear and vestibular pathology
* Worsening of pain or intolerance in the manual cervical traction test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Change in static posturographic parameters: The center of pressure (CoP) movement: sway area | The CoP sway area assessment is done just before the intervention and 5 minutes after.
  The CoP sway area (cm2) correspond to the the area which encloses the data points of the trajectory in relation with the body movement. The CoP sway area is assessed in two conditions (with open then closed eyes)
Change in static posturographic parameters: The CoP displacement amplitude | The CoP displacement amplitude assessment is done just before the intervention and 5 minutes after.
  The CoP displacement amplitude (cm) in the anterior-posterior and medial-lateral trajectory correspond to the amount of body movement during a certain time interval in both trajectories. The CoP displacement amplitude is assessed in two conditions (with open then closed eyes)
Change in static posturographic parameters: The Cop velocity | The Cop velocity assessment is done just before the intervention and 5 minutes after.
  The Cop velocity (cm/s) correspond to the velocity of movement of the body. The CoP velocity is assessed in two conditions (with open then closed eyes)
Change in static posturographic parameters: The Romberg quotient | The Romberg quotient assessment is done just before the intervention and 5 minutes after.
  The Romberg quotient correpond to the Ratio between Closed and Open Eyes Values of the previous parameters.
Change in static posturographic parameters: CoP position | The CoP position assessment is done just before the intervention and 5 minutes after.
  The CoP position correspond to the location side in the frontal plan (left or right) and in the sagittal plan (anterior or posterior). The CoP position is assessed in two conditions (with open then closed eyes)

SECONDARY OUTCOMES:
Change in pain intensity | The pain assessement is done just before the intervention and 5 minutes after
  The pain is assessed using a visual analog scale(VAS) /100 mm (minimum 0 mm and maximum 100 mm). The higher the score the worse the patient's pain.
Change in grip strength (Kg) | The measure is done just before the intervention and 5 minutes after
  The grip strength is measured using Jamar Hydraulic Hand Dynamometer

OTHER OUTCOMES:
The Brief Best test | The test is performed only once at baseline in each patient: before the Effective Traction in the Arm EffectiveTraction/ShamTraction and before the Sham Traction in the Arm ShamTraction/EffectiveTraction.
  Clinical test to assess the balance capacity during standing and walking.
Neck Disability Index (NDI) | The questionnaire is administered only once at baseline in each patient: before the Effective Traction in the Arm EffectiveTraction/ShamTraction and before the Sham Traction in the Arm ShamTraction/EffectiveTraction.
  A self-administered questionnaire used to assess the self-rated disability. It contains 10 sections scored from 0 to 5 each. The total score range from 0 to 50. The higher the score the higher the patient's level of disability.
Hospital Anxiety and Depression scale | The scale is administered only once at baseline in each patient: before the Effective Traction in the Arm EffectiveTraction/ShamTraction and before the Sham Traction in the Arm ShamTraction/EffectiveTraction.
  A scale used to determine the level of anxiety and depression in patients. The questionnaire comprises seven questions for anxiety and seven questions for depression. Each response to a question is scored from 0 to 3. The total score for anxiety and depression separately range from 0 to 21. The higher the score the more sever the patient's anxiety and depression status.
The short form (36) health survey: SF-36 | The questionnaire is administered only once at baseline in each patient: before the Effective Traction in the Arm EffectiveTraction/ShamTraction and before the Sham Traction in the Arm ShamTraction/EffectiveTraction.
  A questionnaire used to assess patient's health status (Quality of life). It yields an 8-scale profile of functional health and well-being scores: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), mental health (MH), and one single item scale on health transition. Score ranges from 0 to 100, with higher score indicating higher level of function and/or better health and lower score indicating lower level of function and/or bad health.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Medicine and rehabilitation Department, Monastir, Tunisia